CLINICAL TRIAL: NCT05571683
Title: Comparison of Cerebral Oxymeter and End Tidal Carbondioxide Values Under Surgical Drapes in Patients With and Without Past COVID-19 Infection Undergoing Cataract Operation
Brief Title: Cerebral Oxymeter and End Tidal Carbondioxide Values Under Surgical Drapes With and Without Past COVID-19 Infection
Status: Completed | Type: Observational
Sponsor: Duzce University (Other)
Responsible Party: Principal Investigator, Özlem Ersoy Karka, Assistant Professor, Duzce University
Other Study IDs: drozlemersoy1
Record Dates: First submitted 2022-10-05; First posted 2022-10-07 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Cataract Extraction; Anesthesia, Local; Optic Nerve Sheath
Keywords: cataract extraction; Anesthesia, Local; optic nerve sheath; carbon dioxide; cerebral oxygen saturation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- recovered from covid-19, 2 l/min oxygen support: 20 patients, who recovered from COVID-19 will be supported with 2 l/min oxygen during the operation under the drapes. Electrocardiography, pulse oximetry, non-invasive blood pressure, end-tidal carbon dioxide and cerebral oximetry will be monitored and optic nerve sheath diameter will be measured before and after surgical procedure. All measurements except optic nerve sheath diameter will be recorded and repeated at 5 minute intervals throughout the operation.
  Interventions: Other: oxygen support
- no covid anamnese, 2 l/min oxygen support: 20 patients with no COVID-19 anamnese will be supported with 2 l/min oxygen during the operation under the drapes. Electrocardiography, pulse oximetry, non-invasive blood pressure, end-tidal carbon dioxide and cerebral oximetry will be monitored and optic nerve sheath diameter will be measured before and after surgical procedure. All measurements except optic nerve sheath diameter will be recorded and repeated at 5 minute intervals throughout the operation.
  Interventions: Other: oxygen support
- recovered from covid-19, 4 l/min oxygen support: 20 patients, who recovered from COVID-19 will be supported with 4 l/min oxygen during the operation under the drapes. Electrocardiography, pulse oximetry, non-invasive blood pressure, end-tidal carbon dioxide and cerebral oximetry will be monitored and optic nerve sheath diameter will be measured before and after surgical procedure. All measurements except optic nerve sheath diameter will be recorded and repeated at 5 minute intervals throughout the operation.
  Interventions: Other: oxygen support
- no covid anamnese, 4 l/min oxygen support: 20 patients with no COVID-19 anamnese will be supported with 4 l/min oxygen during the operation under the drapes. Electrocardiography, pulse oximetry, non-invasive blood pressure, end-tidal carbon dioxide and cerebral oximetry will be monitored and optic nerve sheath diameter will be measured before and after surgical procedure. All measurements except optic nerve sheath diameter will be recorded and repeated at 5 minute intervals throughout the operation.
  Interventions: Other: oxygen support

INTERVENTIONS:
Other: oxygen support — 40 patients (2 arms) will be supported with 2 l/min oxygen and the other 2 arms (40 patients) will be supported with 4 l/min oxygen under the surgical drapes.

SUMMARY:
Today, phacoemulsification has become the most commonly applied method in the treatment of cataract, which is considered as a public health problem. Since the eyelid margins can be a source for pathogens in phacoemulsification surgery draping after skin sterilization is applied to remove the eyelashes from the operation area. Since surgical drapes are airtight, carbon dioxide (CO2) accumulation occurs under the drape in patients under local anesthesia. During the operation, if the end tidal CO2 pressure value rises, this can lead to hyperventilation and tachycardia and also increase the intraocular pressure which is undesirable in eye surgery. In our study, in order to observe and compare undesirable conditions, regional tissue oxygenation saturation (rSO2) will be determined non-invasively with Transcutaneous Near Infrared Spectroscopy (NIRS) technology , which allows real-time monitoring. Changes in the partial pressure of carbon dioxide (PaCO2) are strongly vaso-active, resulting in changes in cerebral blood volume and hence intracranial pressure.

As the optic nerve sheath is an extension of the brain dura mater, the diameter of the sheath expands in case of increased intracranial pressure. Evaluation of the optic nerve sheath with ultrasound allows us to obtain information about intracranial pressure. For optic nerve sheath diameter, measurements above 5.0 mm in adult patients are generally considered as increased intracranial pressure.

COVID-19 is a global epidemic caused by SARS-CoV-2 that we are still fighting. Although it is a multisystemic disease, it is important in terms of its effects on pulmonary function and the continuity of pulmonary symptoms and findings after this disease has been overcome.

In our study, End-Tidal CO2 and cerebral oximetry (NIRS) values will be determined and compared between the groups that received 2lt/min and 4lt/min nasal oxygen support during cataract surgery performed using draping under local anesthesia in patients who had COVID-19, recovered and never had. It was aimed to evaluate and compare the values of optic nerve sheath diameter increase.

DETAILED DESCRIPTION:
After the patients who meet the specified criteria are informed about the study, the volunteers who agreed to participate and signed informed consent will be included in the study.

After all volunteers are taken to the operation room, vascular access will be established, electrocardiography, pulse oximetry, non-invasive blood pressure, end-tidal carbon dioxide and cerebral oximetry (with the neck in the supine position in the neutral position and 2 probes placed on the forehead) are monitored without any medication (Figure 1). The optic nerve sheath diameter will be measured by the ultrasonography device in the inventory of the Department of Anesthesiology and Reanimation by the researchers, basal heart rate (CTA), peripheral oxygen saturation (SpO2), systolic (SBP) and diastolic blood pressure (DBP), end- Tidal carbon dioxide (ETCO2), cerebral oxygen saturation (SO) values will be recorded. All measurements except optic nerve sheath diameter will be recorded and repeated at 5 minute intervals throughout the operation. During this time, no drugs or invasive methods will be used.

During the operation, the volunteers in both groups will be randomly divided into 2 subgroups and 2L/min and 4 L/min nasal oxygen support will be provided. At the end of the operation, the ultrasonographic optic nerve sheath diameter measurement will be repeated immediately after the dressing is removed.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18 who will undergo cataract surgery, who are in I, II and III risk groups according to the American Society of Anesthesiologists (ASA) classification

Exclusion Criteria:

* Patients for whom Intensive Care Unit (ICU) indication is prescribed
* Chronic obstructive pulmonary disease
* Past coronary arterial by-pass graft history
* Hemoglobinopathies
* Neurodegenerative diseases

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 80 patients who will undergo phacoemulsification surgery under local anesthesia will be included in the study.
  40 of the patients will be individuals who have had Covid-19 infection and recovered, and 40 will be individuals who have not had Covid-19 infection.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2022-06-06 (Actual); Primary Completion 2023-12-16 (Actual); Study Completion 2023-12-16 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the end tidal carbon dioxide values | End tidal carbondioxide values will be measured continously during the operation and recorded in every 5 minutes from the draping to the end of the operation.
  End tidal carbondioxide values will be measured continously during the operation with a capnograph device via nasal cannula non-invasively and recorded.
Change from baseline in the cerebral oxygenisation values | Cerebral oxygenisation values will be measured continously during the operation and recorded in every 5 minutes from the draping to the end of the operation.
  Cerebral oxygenisation values will be measured continously during the operation with a transcutaneous near infrared spectroscope device (NIRS) via a transcutaneous probe placed on the frontal bone non-invasively and recorded.
Change from baseline in the optic nerve sheath diameter | 2 times, once before acceptance in the operation room, and secondly on the end of the operation before undraping.
  The optic nerve sheath diameter will be measured ultrasonographically by the same experienced researcher before and on the end of the operation.

CONTACTS AND LOCATIONS:
Overall Officials: Özlem Ersoy Karka, Principal Investigator — Düzce University Faculty of Medicine
Locations (1):
- Duzce University Faculty of Medicine, Düzce, Düzce, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No